CLINICAL TRIAL: NCT05782569
Title: Serial Lung Ultrasound in Predicting the Need for Surfactant and Respiratory Course in Preterm Infants - Observational Study (SLURP)
Brief Title: Serial Lung Ultrasound Predicting Need for Surfactant and Respiratory Course in Preterm Infants Observational Study
Acronym: SLURP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PRENET 2297
Record Dates: First submitted 2023-01-25; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: Infant, Premature
Keywords: Babies born under 34 weeks; Risk of developing lung problems after birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Babies born early (under 34 weeks) are at risk of developing lung problems after birth. A major reason for this is that the lungs are not fully developed (lung immaturity). One of the important components not yet produced by the lungs is the surfactant, which allows premature babies to breathe without much effort. Very often babies born early need some help with their breathing and also need surfactant. Surfactant is administered through a breathing tube which is placed into the baby's airway. It is important that surfactant is administered early after birth when the baby cannot produce it. Early administration of surfactant provides better clinical outcomes.

Currently the decision to give surfactant is based on clinical parameters such as the level of oxygen that your baby requires. Current strategy of waiting for the baby to reach certain oxygen level, may delay in administering surfactant. But recent scientific data from other countries suggest that ultrasound of the chest/lungs can predict early which babies would need surfactant. This would help us to administer surfactant earlier and improve their respiratory outcome. In this study, we want to confirm the value of chest/Lung ultrasound (LU) to predict the need for surfactant in UK population. As a part of the study, we will perform early LU and serial LU in the first few days of life. In this current study, LU images will only be recorded and not used for clinical management.

DETAILED DESCRIPTION:
Participant group for the study: Babies born under 34 weeks with a risk of developing lung problems after birth.

This study is an observational study to confirm the value of chest/Lung ultrasound (LU) to predict the need for surfactant in UK newborn population. As a part of the study, the investigators will perform early LU and serial LU in the first few days of life.

The investigators will perform the first LU within 3 hours of admission. A Second LU will then be taken at 3-6 hours after surfactant administration (if the baby receives surfactant) or at 6-12 hours of life (if the baby continues to be on Non-invasive respiratory support). A third LU is then taken on Day 2 (12-24 hours after the second LU) and a fourth LU on Day 3 (12-24 hours after the third LU). Then the investigators will carry out additional clinical data collection at hospital discharge.

Ultrasound is a common procedure carried out in newborn population. The scan should not take more than 3 to 5 minutes. All other data would be obtained from patient notes and databases.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≤34 weeks based on last menstrual period or ultrasound dating.
2. Non-invasive respiratory support or low flow oxygen needing neonatal unit admission

Exclusion Criteria:

1. Received surfactant before first LU (<3hrs of life).
2. Major congenital malformations including congenital lung disease and congenital heart disease as ascertained by the medical team.
3. Infants receiving delivery room surfactant or required intubation shortly after admission.
4. Infants diagnosed with pneumothorax needing needle or chest tube drainage

Ages: 23 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Recruiting the neonatal (Newborn) population. Currently there is no definite way of identifying which infant would need surfactant so this research would study study the value of lung ultrasound in predicting which infant would benefit from surfactant
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Value of chest/Lung ultrasound (LU) to predict the need for surfactant in preterm population. | 3 hours of age
  Lung ultrasound scores within the first 3 hours of life to predict the need for 1st Dose of surfactant

REFERENCES:
- [Derived] Loganathan PK, Meau-Petit V, Bhojnagarwala B, Nair V, Holmes J, Occhipinti A, Montasser M. Serial lung ultrasound in predicting the need for surfactant and respiratory course in preterm infants-multicentre observational study (SLURP). Eur J Pediatr. 2025 May 23;184(6):356. doi: 10.1007/s00431-025-06185-7. PMID 40407825